CLINICAL TRIAL: NCT00746538
Title: Quality of Life in Patients With Unresectable Hilar Cholangiocarcinoma on Palliative Metallic Stent Versus Plastic Stent: A Randomized Control Trial
Brief Title: Quality of Life in Patients With Unresectable Hilar Cholangiocarcinoma on Palliative Metallic Stent Versus Plastic Stent
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Worrarat Kongkasame, Department of Medice. Faculty of Medicine. Khonkaen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HE500636(subproject); HE5OO636(sub)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-07

CONDITIONS: Unresectable Hilar Cholangiocarcinoma
Keywords: Hilar cholangiocarcinoma; biliary stent; plastic stent; metallic stent; quality of life
MeSH Terms: conditions — Klatskin Tumor | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): metallic stent group
  Interventions: Device: biliary stent
- 2 (Active Comparator): plastic stent group
  Interventions: Device: biliary stent

INTERVENTIONS:
Device: biliary stent — Metallic stent of plastic stent was inserted into right or left hepatic duct which was planed before intervention using CT scan or MRCP
  Other Names: Self expandable metallic stent; Amsterdam type plastic stent

SUMMARY:
The purpose of this study is to compare the quality of life in patients with unresectable hilar cholangiocarcinoma on palliative metallic stent versus plastic Stent.

DETAILED DESCRIPTION:
In the patient with unresectable hilar cholangiocarcinoma,palliative biliary stent is the one way to help him.

The aim of palliative treatment is to improve quality of life and relief symptom,or sometime ,extended survival rate.

There are two types of biliary stent:

1. plastic stent made from polyethylene or polytetrafluoroethylene
2. metalic stent braided in the form of a tubular mesh from surgical-grade stainless steel alloy and designed to expand to a maximum diameter of 10mm.

The main drawback of plastic stent is relatively high occlusion rate, but its advantage is the lower cost.

In the reasons of higher occlusion rate , the lower cost of plastic stent versus metallic stent that should be stent exchange when occluded, so we would to know about quality of life in both group.

ELIGIBILITY:
Inclusion Criteria:

* All patient with diagnosis of hilar cholangiocarcinoma and/or radiological diagnosis
* Patient considered having an unresectable tumor or unfit of operation because of advanced age or medical illness

Exclusion Criteria:

* Patient with ASA 4 or 5
* Patient who inability to comply with follow up
* Patient refused to join the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-03 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
To assessment of the quality of life of patient with unresectable hilar cholangiocarcinoma after palliative biliary stent. | 2-4 weeks

SECONDARY OUTCOMES:
To assessment of early and late complication after palliative stent. | After stent insertion for sixth month and one year or until patients were expired
Survival rate at sixth month and one year. | After stent insertion for sixth month and one year or until patients were expired

CONTACTS AND LOCATIONS:
Overall Officials: Worrarat Kongkasame, MD, Principal Investigator — Department of Medicine.Faculty of Medicine .KhonKaen University
Locations (1):
- Srinagarind Hospital.KhonKaen University., Muang, KhonKaen, Thailand

REFERENCES:
- [Result] De Palma GD, Pezzullo A, Rega M, Persico M, Patrone F, Mastantuono L, Persico G. Unilateral placement of metallic stents for malignant hilar obstruction: a prospective study. Gastrointest Endosc. 2003 Jul;58(1):50-3. doi: 10.1067/mge.2003.310. PMID 12838220
- See also: Research affairs.Faculty of Medicine.KhonKaen University — http://www.md.kku.ac.th/research/index.php?